CLINICAL TRIAL: NCT03517384
Title: Feasibility Pilot Study of Internet-based CBT for Body Dysmorphic Disorder With Global Recruitment
Brief Title: Feasibility Pilot Study of Internet-based Cognitive Behavioral Therapy (CBT) for Body Dysmorphic Disorder With Global Recruitment
Acronym: BDD-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Massachusetts General Hospital (Other); Hofstra University (Other)
Responsible Party: Principal Investigator, Christian Rück, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDD-GLOBAL
Record Dates: First submitted 2018-04-10; First posted 2018-05-07 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Body Dysmorphic Disorders
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I-CBT for Body Dysmorphic Disorder (Experimental): All participants will receive our Internet-Cognitive Behavioral Therapy treatment for Body Dysmorphic Disorder.
  Interventions: Behavioral: I-CBT for Body Dysmorphic Disorder

INTERVENTIONS:
Behavioral: I-CBT for Body Dysmorphic Disorder — The current intervention, is a therapist guided, Internet Cognitive Behavioral Therapy treatment for Body Dysmporhic Disorder which consists of 8 treatment modules administered over the course of 12 weeks.
  Other Names: BDD-NET

SUMMARY:
The aim of the study is to study an english-language version of BDD-NET (Enander, et al., 2014; Enander, et al., 2016), an internet-based treatment for Body Dysmorphic Disorder, on a globally recruited sample. This is an uncontrolled pilot study where a within-subjects repeated measures design was used to assess the feasibility of conducting all aspects of the study remotely, including recruitment, assessment, and treatment delivery.

ELIGIBILITY:
Inclusion Criteria:

* Current outpatient status (not currently admitted for inpatient care)
* Patient is fluent in English
* Patient has regular access to a computer with an Internet connection
* Patient has adequate skills to use the Internet effectively.
* Patient provides informed consent (both verbal, and click yes to consent on secure web page)
* Patient is 18 years of age or older (able to provide government issued photo ID)
* Patient has primary diagnosis of DSM-5 Body Dysmorphic Disorder, (determined using the SCID-5 module "G" which assesses diagnostic criteria on obsessive compulsive spectrum disorders)
* score ≥ 4 on the Body Dysmorphic Disorder Questionnaire (BDDQ),
* score ≥ 9 on the Dysmorphic Concern Questionnaire (DCQ)
* score ≥ 20 on the Body Dysmorphic Disorder Modification of the Yale Brown Obsessive Compulsive Scale (BDD-YBOCS).

Exclusion Criteria:

* Patient received Cognitive Behavior Therapy for Body Dysmporphic Disorder in the 12 months preceding treatment
* Patient changed psychotropic medications within the 12 weeks before treatment
* Patient receiving other ongoing psychotherapy at the time,
* Patient did not have access to a 24 hour psychiatric emergency center
* Patient could not provide an emergency contact person.
* Current substance dependence (assessed with M.I.N.I. 7.0, AUDIT, DUDIT)
* Lifetime bipolar disorder diagnosis (assessed with M.I.N.I. 7.0 and self-report)
* Psychosis present
* Severe depression (assessed with M.I.N.I., MADRS-S score ≥ 35)
* Personality disorder diagnosis (self-report and video-conference diagnostic interview),
* Lifetime history of suicide attempts (self-report) or clinically significant current suicidal ideation (≥ 5 on item 9 of MADRS-S; Columbia Suicide Severity Rating Scale (C-SSRS Lifetime Recent) - Clinical Version: Recent (past month) - Most Severe Ideation score ≥ 4).
* Additionally, eligibility continues to be assessed on an ongoing basis after initial inclusion. The MADRS-S, Appearance Anxiety Questionnaire (AAI), and Adverse Events Questionnaire (AEQ) are administered weekly in order to ensure that the treatment study continues to be a safe and appropriate level of care for participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Symptom Change using the Clinician-rated, Body Dysmporhic Disorder Modification of Yale-Brown Obsessive Compulsive Scale (BDD-YBOCS) | baseline, week 6, post (week 12), 3 month follow-up, 12 month follow-up
  A measure of BDD symptom severity. Scores range from 0-48 with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Structured Clinical Interview for Diagnostic Statistical Manual 5th edition (DSM 5) - Research Version (SCID-5-RV) module G | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  assessment of BDD diagnostic status
Mini-International Neuropsychiatric Interview - version 7.0 (M.I.N.I. 7.0) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  assessment of current major depressive episode and other comorbid anxiety diagnoses
Dysmorphic Concerns Questionnaire (DCQ) | screening, baseline, post (week 12), 3 month follow-up, 12 month follow-up
  used for BDD screening/ measuring dysmorphic concerns. Scores range from 0 to 28 with higher scores indicating higher severity
Appearance Anxiety Inventory (AAI) | screening, baseline, weeks 1-11, post (week 12), 3 month follow-up, 12 month follow-up
  A measure of BDD symptoms. The maximum total score is 40, with higher scores indicating greater frequency of a process
Brown Assessment of Beliefs Scale (BABS) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  Measures conviction and insight regarding beliefs/ obsessions. Scores can range from 0 to 24 with higher scores indicating poorer insight.
Montgomery-Åsberg Depression Rating Scale, self-report (MADRS-S) | screening, baseline, weeks 1-11, post (week 12), 3 month follow-up, 12 month follow-up
  measures depressive symptoms and suicidal ideation. Scores range from 0-54 with higher scores indicating higher severity.
Skin-Picking Scale - Revised (SPS-R) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  Measures skin picking severity. Scores range from 0 to 32 with higher scores indicating higher severity
Global Assessment of Functioning (GAF) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  A measure of global functioning. Scores range from 0-100 with higher scores indicating better functioning.
Clinical Global Impressions Scale - Severity (CGI-S) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  measures global severity. Scores range from 1-7 with higher scores indicating more severity.
Clinical Global Impressions Scale - Improvement (CGI-I) | post (week 12), 3 month follow-up, 12 month follow-up
  measures global improvement. Scores range from 1-7 with low scores indicating more improvement.
EuroQol - 5 Dimension Questionnaire (EQ-5D) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  Measures quality of life and functioning. Scores range between 0 (dead) and 1 (perfect health).
Sheehan Disability Scale (SDS) | baseline, post (week 12), 3 month follow-up, 12 month follow-up
  The SDS has 3 items measuring functional impairment and disability regarding work/school, social life/leisure, and family life/home responsibilities on a likert scale between 0 (no interference) to 10 (extreme impairment). Two items measure days lost at work/school and days being underproductive at work/school. Items are on a likert scale of 0 (not at all) to 10 (very severe).
Client Satisfaction Inventory (CSI) | weeks 2, 7, and 12 (post)
  Measures participants' satisfaction with treatment. Total raw scores on this measure range 0 to 175 with higher scores indicating higher satisfaction
Working Alliance Inventory - Short Revised (WAI-SR) | weeks 2, 4, 6, 8, 10, and 12 (post)
  Measures working alliance between therapist and patient. Scores range from 0-60 with higher scores indicating better working alliance.
Credibility Scale (Credibility/Expectancy Questionnaire) | baseline, weeks 2, 4, 6, 8, 10, and 12 (post)
  Measures patients' perception of the credibility of treatment and expectations for treatment outcome. Scores range from 0-55 with higher scores indicating better expectations of treatment outcome and higher perceptions that the treatment is credible.
Internet Cognitive Behavioral Therapy -- Exposure and Response Prevention Adherence Scale (ICBT - EX/RP Adherence Scale, modified from the Patient EX/RP Adherence Scale (PEAS)) | weeks 2-11, and week 12 (post)
  Measures patients adherence to treatment. Raw scores range from 0-62 with higher scores indicating more adherence to treatment.
Completion of Core Treatment Modules | Post treatment (Week 12)
  Have participants completed modules 1-5?
Early Termination Checklist | Post treatment (Week 12)
  indicates possible reasons for participants early termination from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enander J, Andersson E, Mataix-Cols D, Lichtenstein L, Alstrom K, Andersson G, Ljotsson B, Ruck C. Therapist guided internet based cognitive behavioural therapy for body dysmorphic disorder: single blind randomised controlled trial. BMJ. 2016 Feb 2;352:i241. doi: 10.1136/bmj.i241. PMID 26837684
- [Background] Enander J, Ivanov VZ, Andersson E, Mataix-Cols D, Ljotsson B, Ruck C. Therapist-guided, Internet-based cognitive-behavioural therapy for body dysmorphic disorder (BDD-NET): a feasibility study. BMJ Open. 2014 Sep 25;4(9):e005923. doi: 10.1136/bmjopen-2014-005923. PMID 25256187
- [Result] Gentile AJ, La Lima C, Flygare O, Enander J, Wilhelm S, Mataix-Cols D, Ruck C. Internet-based, therapist-guided, cognitive-behavioural therapy for body dysmorphic disorder with global eligibility for inclusion: an uncontrolled pilot study. BMJ Open. 2019 Mar 23;9(3):e024693. doi: 10.1136/bmjopen-2018-024693. PMID 30904854